CLINICAL TRIAL: NCT00023127
Title: Reducing Indoor Allergen Exposures in Northern Manhattan and the South Bronx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9142-CP-001
Record Dates: First submitted 2001-08-22; First posted 2001-08-24 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Asthma; Allergy
Keywords: Asthma; Allergen; Cockroach
MeSH Terms: conditions — Asthma; Hypersensitivity

INTERVENTIONS:
Procedure: Integrated Pest Management

SUMMARY:
Controlled trial of an intervention to reduce indoor exposures to cockroach allergens among asthmatic children in NYC.

ELIGIBILITY:
Ages 6-18

Doctor-diagnosed asthma

Skin-test reactivity to cockroach antigen

Daily cockroach sitings in home

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (1):
- Mailman School of Public Health at Columbia University, New York, New York, United States